CLINICAL TRIAL: NCT03765528
Title: Impact of Prescription Quality, Infection Control and Antimicrobial Stewardship on Gut Microbiota Domination by Healthcare-Associated Pathogens
Acronym: PILGRIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Collaborators: University Hospital of North Norway (Other); Karolinska Institutet (Other); Rabin Medical Center (Other); University of Latvia (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Haukeland University Hospital (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); Goethe University (Other)
Responsible Party: Principal Investigator, Dr. med. Jörg Janne Vehreschild, Professor, University Hospital of Cologne
Other Study IDs: PILGRIM
Record Dates: First submitted 2018-11-16; First posted 2018-12-05 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Patients at High Risk of Antibacterial Treatment Upon Admission
Keywords: Clostridium difficile; Extended-Spectrum β-Lactamase producing Enterobacteriaceae; Vancomycin-resistant enterococci; Antimicrobial resistance; Microbiome; Nosocomial infection; Antimicrobial Stewardship; Infection Control
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extended-spectrum beta-lactamase producing Enterobacteriaceae (EPE), vancomycin-resistant enterococci (VRE) and Clostridium difficile have become a major threat to hospitalised patients worldwide. We hypothesize that receiving inappropriate antibacterial treatment places patients at high risk of intestinal domination and subsequent infection by these bacteria. Further analyses will address cost-effectiveness of specific interventions, behavioural analyses of the decision process leading to inappropriate antibacterial treatment, and the rate of undetected colonization with EPE/VRE/C. difficile on admission.

DETAILED DESCRIPTION:
The prevalence of antimicrobial resistant pathogens has dramatically increased among hospitalised patients worldwide. While various management strategies have effectively reduced the burden caused by methicillin-resistant Staphylococcus aureus, resistant pathogens with a preference towards intestinal colonization are currently on the rise. E.g., vancomycin-resistant enterococci (VRE) and extended-spectrum beta-lactamase producing Enterobacteriaceae (EPE) now constitute a significant threat to hospitalised patients worldwide, as infections due to these organisms require prolonged treatments and result in inferior outcomes. Similarly, the burden of disease caused by Clostridium difficile infection (CDI), the main cause of healthcare-associated infectious diarrhoea, has increased driven by the emergence of hypervirulent strains such as ribotypes 027 and 078. Molecular studies have demonstrated that increased population-wide exposure to broad-spectrum antibacterials is a crucial step in the initiation of outbreaks by selection and expansion of resistant C. difficile.

This is a comprehensive, multinational, multi-centre clinical study aiming to assess the impact of inappropriate antibacterial prescription on intestinal domination by EPE or VRE or infection with C. difficile. To achieve this goal, the study will closely follow the progression from first acquisition of drug-resistant organisms to infection with these bacteria at an individual patient level.

In this study, we will establish the sequence and factors involved in acquisition, colonization, selective pressure, bacterial overgrowth/domination/ and infection for EPE, VRE and C. difficile. We hypothesize that IC (Infection Control; prevention of pathogen acquisition) and AMS (Antimicrobial Stewardship; prevention of clonal expansion) measures leading to a higher share of appropriate anti-infective use are effective strategies to prevent this development. The study programme will allow an accurate estimation of the preventable share of healthcare-acquired colonization and infection by VRE, EPE, and C. difficile.

No direct interventions will be performed with study patients. Instead, study centres will assess quality indicators for implementation of IC and AMS measures by active observation and aggregation of data. Patients fulfilling all inclusion- and no exclusion criteria will be asked for their consent to be recruited prospectively into a cohort study. During the observational phase, participants will be monitored for receipt of antibacterial treatment and regular stool samples will be obtained and stored. An interdisciplinary, international AMS Board will comprehensively assess antibiotic treatment via review by a panel of experts. After the observation is completed, stool samples will be batch-tested for intestinal domination by the target pathogens of this study. Statistical analyses will be performed to investigate an association between inappropriate antibiotic use as opposed to appropriate or no antibiotic use and intestinal domination. If domination is detected, further analyses for phenotype, quantity, resistance, and molecular biology will be performed. Finally, the baseline sample will be tested for presence of the dominant species to understand the source of the pathogen, i.e. nosocomial versus outpatient acquisition.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Planned treatment or high likelihood of any systemic antibacterial treatment except trimethoprim/sulfamethoxazole within the next 10 days for a duration of ≥ 5 days
3. Patients able to provide a stool sample before or within 4 hours of receiving first antibiotic dosage
4. Written informed consent provided prior to inclusion

Exclusion Criteria:

1. Patients who have received courses of systemic antibacterials for 7 days or more within the past two months
2. Patients having received any antibacterial compound other than trimethoprim/sulfamethoxazole within 14 days prior to study enrolment except first antibiotic dosage within 4 hours prior enrolment
3. Patients with diarrhea at enrolment (≥3 unformed bowel movements within 24h)
4. Patients with a stoma (jejunostomy, ileostomy, or colostomy) at time of inclusion
5. Patients on enteral (tube fed or PEG) or parenteral nutrition
6. Patient with any social or logistical condition which in the opinion of the investigator may interfere with the conduct of the study, such as incapacity to well understand, not willing to collaborate, or cannot easily be contacted after discharge
7. Patients exclusively treated as outpatients without prior hospital admission
8. Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients at high risk of receiving antibiotic treatment during their hospital stay will be screened for study eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Impact of inappropriate antibacterial prescription on intestinal microbiota domination by healthcare associated pathogens | up to 6 - 36 weeks
  The differential impact of inappropriate antibacterial prescription compared to adequate or no antibacterial prescription on intestinal microbiota domination by EPE or VRE or infection with C. difficile measured by analysing stool samples.

SECONDARY OUTCOMES:
Time-point of Intestinal Colonization | Baseline and up to 6 - 36 weeks
  Determination of the rate of in-hospital vs. pre-admission intestinal colonization with EPE, VRE, and/or C. difficile measured by analysing stool samples.
Time-point of Intestinal Domination | Baseline and up to 6 - 36 weeks
  Determination of the rate of in-hospital vs. pre-admission intestinal domination with EPE, VRE, and/or C. difficile measured by analysing stool samples.
Inter-rater reliability of AMS specialists | After complete documentation of each patient case (follow-up for 6-36 weeks) followed by completed ratings of AMS specialists
  Determination of the inter-rater reliability of interdisciplinary AMS specialists rating antibacterial prescription appropriateness.
Rationale for antibacterial prescription habits assessed by performing qualitative interviews with prescribing physicians | After complete documentation of patient case (follow-up for 6-36 weeks) through study completion
  Identification of behavioral determinants and knowledge gaps leading to inappropriate antibacterial prescriptions by interviewing approximately 50 prescribing physicians.
Correlation of prescription and AMS implementation | Baseline, 12 months, 24 months
  Assessment of the correlation of appropriate antibacterial prescription with quality indicators of AMS implementation
Identification of risk factors responsible for disrupting the intestinal microbiota | Baseline and weekly up to 6 - 36 weeks of follow-up
  Identification of risk factors for colonization, intestinal domination, and infection by EPE, VRE and C. difficile, including comorbidities and drugs known to disrupt the intestinal microbiota, and high-risk bacterial clones prone to dominate the microbiota due to high fitness. Assessment by analysing stool samples and documented data.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Janne Vehreschild, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No